CLINICAL TRIAL: NCT07061041
Title: Comparison of the Effects of Static Stretching and Full Range of Motion Strength Training on Posterior Band Flexibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Principal Investigator, Michał Kaczorowski, Laboratory Assistant, Józef Piłsudski University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SKE.0030.59.2025
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Flexibility; Strength Training Effects; Static Stretching
Keywords: flexibility; static streching; minimal-dose; hamstring flexibility
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Only tests were performed in the group, no intervention was introduced
- Streching group (Experimental): The group performed one training session per week consisting of 2 sets of 60 seconds of static stretching
  Interventions: Other: Streching group
- Strength training group (Experimental): The group will perform one workout per week consisting of 3 series of the "Romanian deadlift" exercise of 10 repetitions. Each repetition will be performed at a specific pace - 3s in eccentric contraction and 1s in concentric contraction. The aforementioned exercise, the Romanian deadlift, will be performed by the subjects on a platform (elevation) in order to achieve maximum range of motion.
  Interventions: Other: Strength training

INTERVENTIONS:
Other: Strength training — The group will perform one workout per week consisting of 3 series of the "Romanian deadlift" exercise of 10 repetitions. Each repetition will be performed at a specific pace - 3s in eccentric contraction and 1s in concentric contraction. The aforementioned exercise, the Romanian deadlift, will be performed by the subjects on a platform (elevation) in order to achieve maximum range of motion.
  Arms: Strength training group
Other: Streching group — The group performed one training session per week consisting of 2 sets of 60 seconds of static stretching
  Arms: Streching group

SUMMARY:
The study will be conducted in 2025. The methods used in the study are non-invasive methods. One study group will perform 2 series of static stretching of the posterior band once a week. The stretching time in each series will be 60s, and the duration of the intervention will be 6 weeks. The test subjects will maintain a maximum prone position with their knee joints straight for a specified period of time during the stretching. The second study group will perform full range of motion strength training in the form of 3 series of 10 repetitions of the Romanian Deadlift (RDL) once a week, with the intervention duration also being 6 weeks. Prior to the start of the study, participants will undergo a toe-to-floor test to assess posterior band flexibility. The test will be repeated again after the intervention.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years,
* No lower limb injuries, no spinal injuries and no craniocerebral injuries in the last 6 months,
* No lower limb surgeries, no spinal surgeries and no central nervous system surgeries in the last 6 months,

Exclusion Criteria:

* Age under 18 years
* Injuries to the lower limbs, spine or craniocerebral injuries within the last 6 months,
* Surgical procedures to the lower limbs, spine or surgical procedures to the central nervous system within the last 6 months,

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
Flexibility | From registration to completion of the study, the duration is up to 8 weeks
  Flexibility was assessed using a modified stand-and-reach test. The participants stood with their feet shoulder-width apart and knees fully extended, then performed a forward bend, reaching as far as possible while maintaining straight legs. To measure the extent of their reach, a custom-built box was used. The box had the following dimensions: a length of 40 cm, a width of 45 cm, and a height of 35 cm. Each participant performed the test once. The same test was repeated after the 6-week intervention period to determine any improvements in flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Józef Piłsudski Academy of Physical Education in Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shadmehr A, Hadian MR, Naiemi SS, Jalaie S. Hamstring flexibility in young women following passive stretch and muscle energy technique. J Back Musculoskelet Rehabil. 2009;22(3):143-8. doi: 10.3233/BMR-2009-0227. PMID 20023343
- [Background] Zhao S, Robertson DD, Wang G, Whiting B, Bae KT. X-ray CT metal artifact reduction using wavelets: an application for imaging total hip prostheses. IEEE Trans Med Imaging. 2000 Dec;19(12):1238-47. doi: 10.1109/42.897816. PMID 11212372